CLINICAL TRIAL: NCT00139035
Title: Effects of Cyclosporine A on Pancreatic Insulin Secretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CsA-Dialysis 2004-004488-3
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Renal Failure
Keywords: glucose intolerance; insulin; microvascular function; genotyping; CYP3A5; pharmacokinetics; renal transplantation
MeSH Terms: conditions — Kidney Failure, Chronic; Glucose Intolerance; Insulin Resistance | interventions — Cyclosporine

INTERVENTIONS:
Drug: cyclosporine A

SUMMARY:
Our primary aim is to investigate if cyclosporine A reduces insulin secretion.

DETAILED DESCRIPTION:
Our primary aim is to investigate if cyclosporine A may reduce insulin secretion by 20% or more. In order to get cyclosporine A naïve patients we will perform this investigation in dialysis patients on the waiting list for a renal transplantation. In addition we will investigate if also the peripheral insulin sensitivity and endothelia function is affected by cyclosporine A treatment in these patients. Since these patients will be treated with cyclosporine A we will also measure cyclosporine pharmacokinetics at the time of investigation and repeat this investigation at the time of the first week following transplantation in order to evaluate if a pretransplant cyclosporine dose can be of value in predefining the dose to be used at the time of transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Renal failure patients on dialysis which is planned to receive a renal transplant

Exclusion Criteria:

* Age below 18 years or above 75 years
* Pregnancy
* Breast feeding mothers
* Diabetes mellitus /WHO criteria)
* Dialysis treatment less than 2 months
* Serious coronary heart disease
* Unstable angina pectoris
* Recent acute infarction (less than 3 months)
* Non-compensated heart failure
* Simultaneous treatment with glucocorticosteroids (e.g. prednisolone, dexamethasone), diltiazem, verapamil, erythromycin, clarithromycin, telithromycin, rifampicin, fluconazole, itraconazole, ketoconazole, voriconazole, indinavir, nelfinavir, ritonavir, nefazodone, bosentan, carbamazepine, St. John's worth, grapefruit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2005-04; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Insulin secretion

SECONDARY OUTCOMES:
Peripheral insulin sensitivity
Endothelial function
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, MSc, Study Director — University of Oslo
Locations (1):
- Rikshospitalet, Section of Nephrology, Oslo, Oslo County, Norway